CLINICAL TRIAL: NCT05268770
Title: The Role of Inflammation in the Pathogenesis of Tinnitus
Brief Title: Inflammation in Tinnitus
Acronym: INFLATIN
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 202200148
Record Dates: First submitted 2022-02-24; First posted 2022-03-07 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Tinnitus, Subjective; Tinnitus; Inflammation
MeSH Terms: conditions — Tinnitus; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tinnitus patients with good hearing
- Healthy controls with good hearing

SUMMARY:
Rationale: Tinnitus is the perception of sound without an external source. In the past decade, inflammation has been implicated in the pathophysiology of tinnitus. In animal models of tinnitus, the expression of proinflammatory cytokines Tumor Necrosis Factor-α (TNF-α) and interleukine-1β (IL-1β) was increased throughout the whole auditory tract. Only two studies evaluated cytokine concentrations in tinnitus patients. In these studies an increase of IL-6 and decrease of IL-10 have been objectified. However, studies did not include tinnitus patients based on the degree of hearing loss, despite that inflammation has also been implicated in hearing loss. On the other hand, studies about inflammation in hearing loss did not (always) exclude tinnitus. Thus, it remains unclear whether the upregulated cytokine concentrations the studies are specific for tinnitus, and whether potential effects remained unsignificant because the presence of hearing loss is a confounder. Therefore, the aim of this study is to evaluate the presence of inflammation in tinnitus patients with normal hearing.

Objective: The main objective is to evaluate the presence of inflammation in blood samples of human subjects with tinnitus and normal hearing, compared to healthy controls. The secondary objective is to evaluate the relation between tinnitus severity and inflammatory marker concentrations.

Study design: This is a cross-sectional study.

Study population: Patients who have been referred to the tinnitus consultation at the outpatient clinic will be asked to participate in this study. For the control group, healthy volunteers will be recruited.

Main study parameters/endpoints: The main study parameter is the disparity in blood cytokine levels between participants with and without tinnitus. Secondary study parameters are the relation between tinnitus severity and blood cytokine concentration, and the difference in complete blood count measures in participants with and without tinnitus.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate in this study, a subject must meet all of the following criteria:
* Adult, aged 18 years or older;
* Hearing threshold: average of 1000kHz, 2000kHz & 4000kHz ≤ 25 dB.
* Anxiety score HADS ≤ 7
* Depression score HADS ≤ 7
* Participant has sufficient mastery of the Dutch language to fill out the questionnaires.
* Psychosocially, mentally, and physically able to fully comply with this protocol.

Exclusion Criteria:

* Objective tinnitus.
* Presence of neurological disease (apart from tinnitus)
* Presence of inflammatory disease, or the use of anti-inflammatory medication.
* Presence or history of a malignancy
* Presence of a disease of the ear (e.g. chronic otitis media, otosclerosis, previous surgery etc).
* Presence of an coagulation disorder
* Presence of a serious psychiatric disorder.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients seeking medical attention at the tinnitus consultation of the otorhinolaryngology department are eligible. Each week, six patients attend the tinnitus consultation. From these patients, we estimate that about a third of the patients meets the inclusion criteria. Additionally, tinnitus patients can be recruited from the tinnitus database of the otorhinolaryngology department. As controls, healthy participants without tinnitus will be included. We expect no difficulties recruiting the planned number of patients from both populations.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Tinnitus vs no tinnitus | September 2022
  Difference in cytokine levels between participants with and without tinnitus

SECONDARY OUTCOMES:
Tinnitus severity | September 2022
  Relation between cytokine levels and tinnitus severity

IPD SHARING:
Plan to Share IPD: No